CLINICAL TRIAL: NCT00889889
Title: Randomized, Double-Blind, Placebo-Controlled Study to Assess the Immunogenicity and Safety of a Cell-Derived Trivalent Subunit Influenza Vaccine in Subjects Aged >= 18 Years and <= 64 Years During Two Consecutive Years.
Brief Title: Immunogenicity and Safety of a Cell-derived Influenza Vaccine in Adults Aged >= 18 and <= 64, Plus Revaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Biologicals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S203.2.004
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-09

CONDITIONS: Influenza
Keywords: Influenza; Phase II; Placebo-controlled
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Cell-Derived Trivalent Subunit Influenza Vaccine
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Cell-Derived Trivalent Subunit Influenza Vaccine — surface antigen, inactivated, prepared in cell cultures
  Arms: 1
Biological: Placebo — Placebo
  Arms: 2

SUMMARY:
Immunogenicity and safety of a cell-derived influenza vaccine in adults aged >= 18 and <= 64 years, plus revaccination

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to give informed consent and able to adhere to all protocol required study procedures.
2. Men and women aged >= 18 and <= 64 years.
3. Being in good health as judged by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria

1. Known to be allergic to constituents of the vaccine.
2. A serious adverse reaction after a previous (influenza) vaccination. Presence of any significant condition that may prohibit inclusion as determined by the investigator.
3. Having received vaccination against influenza or lab confirmed influenza within the previous six months before study vaccination.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1270 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the immunogenicity of the cell-derived subunit vaccine three weeks after vaccination, by applying the FDA requirement for influenza vaccines. | 3 weeks
To assess after the first vaccination the safety and tolerability of the cell-derived subunit vaccine compared to placebo. | 6 months

SECONDARY OUTCOMES:
To assess the long-term immunogenicity (6 months) of the cell-derived subunit vaccine. | 6 months
To assess the immunogenicity of the cell-derived subunit vaccine three weeks after revaccination. | 3 weeks
To assess after the second vaccination the safety and tolerability of the cell-derived subunit vaccine. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanka de Voogd, MD, Study Director — Abbott
Locations (15):
- United States (15):
  - Site Reference ID/Investigator# 45690, Jacksonville, Florida
  - Site Reference ID/Investigator# 45687, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 45697, South Miami, Florida
  - Site Reference ID/Investigator# 45691, Lenexa, Kansas
  - Site Reference ID/Investigator# 45689, Overland Park, Kansas
  - Site Reference ID/Investigator# 45694, Wichita, Kansas
  - Site Reference ID/Investigator# 45682, Lexington, Kentucky
  - Site Reference ID/Investigator# 45684, Kansas City, Missouri
  - Site Reference ID/Investigator# 45685, Omaha, Nebraska
  - Site Reference ID/Investigator# 45686, Las Vegas, Nevada
  - Site Reference ID/Investigator# 45688, Raleigh, North Carolina
  - Site Reference ID/Investigator# 45696, Nashville, Tennessee
  - Site Reference ID/Investigator# 45683, Austin, Texas
  - Site Reference ID/Investigator# 45695, Fort Worth, Texas
  - Site Reference ID/Investigator# 45692, Salt Lake City, Utah